CLINICAL TRIAL: NCT05525520
Title: Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Effects of EP547 in Subjects With Cholestatic Pruritus Due to Primary Biliary Cholangitis or Primary Sclerosing Cholangitis
Brief Title: Study to Evaluate EP547 in Subjects With Cholestatic Pruritus Due to Primary Biliary Cholangitis or Primary Sclerosing Cholangitis
Acronym: PACIFIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Escient Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EP-547-201; 2021-002526-25 (EudraCT Number)
Record Dates: First submitted 2022-08-30; First posted 2022-09-01 (Actual); Results first posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Pruritus
Keywords: Pruritus; Itch; Primary Biliary Cholangitis; Primary Sclerosing Cholangitis; PACIFIC; EP547
MeSH Terms: conditions — Pruritus; Liver Cirrhosis, Biliary; Cholangitis, Sclerosing

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EP547 100 mg (Experimental)
  Interventions: Drug: EP547
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EP547 — Once daily
  Arms: EP547 100 mg
Drug: Placebo — Once daily
  Arms: Placebo

SUMMARY:
This phase 2 trial will evaluate the effects of EP547 in subjects with cholestatic pruritus due to Primary Biliary Cholangitis (PBC) or Primary Sclerosing Cholangitis (PSC)

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80 years
* Documented primary biliary cholangitis (PBC) or primary sclerosing cholangitis (PSC)
* Presence of consistent moderate to severe pruritus
* Use of anti-pruritic and anti-cholestatic (including UDCA and obeticholic acid) medication allowed if meeting additional criteria
* Individuals with concomitant inflammatory bowel disease must meet additional relevant criteria

Exclusion Criteria:

* Pruritus associated with an etiology other than PBC or PSC
* Prior or planned liver transplantation
* Evidence of compensated or decompensated cirrhosis
* Alternative causes of liver disease
* Presence of documented secondary sclerosing cholangitis
* Current evidence of clinically significant high-grade strictures or presence of biliary stent
* History of significant small bowel resection or short bowel syndrome
* Has exclusionary laboratory or biochemical results at Screening

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2022-10-06 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2024-09-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (52):
- United States (21):
  - University of Alabama Birmingham Hospital, Birmingham, Alabama
  - Dignity Health Center for Clinical Research at St. Joseph Hospital, Phoenix, Arizona
  - Southern California Research Center, Coronado, California
  - Science 37, Culver City, California
  - California Liver Research Institute, Pasadena, California
  - University of Miami - Schiff Center for Liver Diseases, Miami, Florida
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Ochsner Medical Center, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - NYU Grossman School of Medicine Gastroenterology and Hepatology, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Gastro Health Research, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - UPMC Center for Liver Disease, Pittsburgh, Pennsylvania
  - The Liver Institute at Methodist Dallas Medical Center, Dallas, Texas
  - Liver Associates of Texas, PA, Houston, Texas
  - Gastro Health & Nutrition, Katy, Texas
  - Digestive & Liver Disease Specialists, Norfolk, Virginia
  - Bon Secours Liver Institute of Virginia, Richmond, Virginia
- Belgium (3):
  - UZ Antwerpen, Antwerp
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
- Canada (4):
  - University of Alberta, Edmonton, Alberta
  - (G.I.R.I.) GI Research Institute, Vancouver, British Columbia
  - Toronto Centre for Liver Disease Toronto General Hospital, Toronto, Ontario
  - Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebeck
- France (6):
  - APHP Avicenne, Bobigny
  - CHU Grenoble- Alpes- Site Nord, Grenoble
  - CHU de Lille, Lille
  - Saint Antoine Hospital, Paris
  - Hospital Rangueil, Toulouse
  - Paul Brousse Hospital, Villejuif
- Israel (4):
  - Carmel Medical Center, Haifa
  - Rambam Medical Center- Keriat Eliezer Family Health Center, Haifa
  - Hadassah Medical Center (Ein-Karem), Jerusalem
  - Chaim Sheba Medical Center, Ramat Gan
- Academic Medical Center- University of Amsterdam, Amsterdam, Netherlands
- Spain (6):
  - Hospital General Universitario Alicante, Alicante
  - Hospital Clinic Barcelona, Barcelona
  - Hospital de Montecelo, Pontevedra
  - Campus Hospital Universitario Virgen del Rocio, Seville
  - La Fe University and Polytechnic Hospital, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- United Kingdom (7):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Glasgow Royal Infirmary, Glasgow
  - King's College Hospital NHS Foundation Trust, London
  - Institute of Cellular Medicine, Newcastle University, Newcastle
  - Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich
  - University of Nottingham - Nottingham Digestive Diseases Centre Biomedical Research Unit, Nottingham
  - University Hospitals Plymouth NHS Trust - Derriford Hospital, Plymouth

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were enrolled at 29 study sites across the United States, United Kingdom, France, Spain, Canada, Israel, Belgium, and the Netherlands.
Groups:
- Placebo 100 mg QD; EP547 100 mg QD: Participants were randomized to receive oral placebo 100 mg QD for 6 weeks in the Double-Blind (DB) Treatment Period. Participants who completed the Double-Blind Treatment Period and were still receiving study drug switched to oral EP547 100 mg QD for 6 weeks in the Open-Label Extension Period.
- EP547 100 mg QD; EP547 100 mg QD: Participants were randomized to receive oral EP547 100 milligrams (mg) once daily (QD) for 6 weeks in the Double-Blind Treatment Period. Participants who completed the Double-Blind Treatment Period and were still receiving study drug received oral EP547 100 mg QD for an additional 6 weeks in the Open-Label Extension Period.
Period: DB Treatment Period (Weeks 1-6)
Arm/Group | Placebo 100 mg QD; EP547 100 mg QD | EP547 100 mg QD; EP547 100 mg QD
Started | 30 | 32
Completed | 29 | 29
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Protocol Violation | 1 | 1
Period: Open-label Extension Period (Weeks 7-12)
Arm/Group | Placebo 100 mg QD; EP547 100 mg QD | EP547 100 mg QD; EP547 100 mg QD
Started | 29 | 29
Completed | 29 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Data are reported for the Full Analysis Set, comprised of all participants who were randomized and took at least 1 dose of randomized study drug. Participants were analyzed according to randomized treatment assignment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo 100 mg QD; EP547 100 mg QD | EP547 100 mg QD; EP547 100 mg QD | Total
Number analyzed (Participants) | 30 | 31 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.6 (12.99) | 51.6 (12.88) | 51.1 (12.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 24 | 48
  Male | 6 | 7 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 10
  Not Hispanic or Latino | 25 | 24 | 49
  Unknown or Not Reported | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 1 | 1
  Black or African American | 3 | 3 | 6
  White | 26 | 25 | 51
  Asian/White | 1 | 0 | 1
  American Indian or Alaska Native/White | 0 | 1 | 1
  North African (Morocco) | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Worst Itch Numeric Rating Scale (WI-NRS) Score up to Week 6
Description: Participants were asked to rate the severity of their worst level of itching in the past 24 hours using the daily WI-NRS, an 11-point scale ranging from 0 (no itching) to 10 (worst itching imaginable). Itching severity scores collected via the WI-NRS have been categorized in the as mild (<4), moderate (≥4 to <7), or severe (≥7). The average WI-NRS score using the daily values from the week before the first dose of study drug (including the WI-NRS score captured on Study Day 1 of dosing) served as the Baseline score. A weekly score was determined based on the average of all available daily scores of the week. Change from Baseline was calculated as the post-Baseline score minus the Baseline score.
Time Frame: Baseline; up to Week 6
Population: Full Analysis Set: all participants who were randomized and took at least 1 dose of randomized study drug. Participants were analyzed according to randomized treatment assignment. Only participants with available data were analyzed. MMRM=mixed effects model for repeated measures.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo 100 mg QD; EP547 100 mg QD | EP547 100 mg QD; EP547 100 mg QD
Number analyzed (Participants) | 27 | 30
scores on a scale | -2.20 (0.445) | -1.75 (0.430)
Statistical Analysis 1: Comparison: Placebo 100 mg QD; EP547 100 mg QD vs EP547 100 mg QD; EP547 100 mg QD; Test type: Equivalence — two-sided equivalence test; p = 0.4577, MMRM; Treatment, type of cholestatic disease, week, and treatment-by-week interaction were fixed effects, and Baseline WI-NRS score was a covariate; Least square mean difference (LSMD) = 0.46, 95% CI 2-sided [-0.77 to 1.68], Standard Error of Mean 0.609 — LSMD=EP547 minus placebo

2. Secondary Outcome: Change From Baseline in the 5-D Itch Scale Total Score at Week 6
Description: The 5-D Itch Scale is a multidimensional (degree, duration, direction, disability, and distribution) questionnaire measuring changes in pruritis. The duration, degree, and direction domain scores range from 1 (no pruritus) to 5 (most severe pruritus). The disability domain includes 4 items assessing itching impact on daily activities: sleep, leisure/social activities, housework/errands, and work/school. Disability domain score=highest score on any of the 4 categories (1 [no pruritis] to 5 [most severe pruritis]). For the distribution domain, 16 body parts are listed to determine the distribution of itching over the last 2 weeks; the number of affected body parts is tallied (potential sum=0-16); the sum is sorted into 5 thresholds: 0-2 is assigned a score of 1; 3-5, a score of 2; 6-10, a score of 3; 11-13, a score of 4; 14-16, a score of 5. Higher scores indicate more severe pruritis. The 5 domain scores are summed to get a total 5-D score: 5 (no pruritus) to 25 (most severe pruritus).
Time Frame: Baseline; Week 6
Population: Full Analysis Set. Only participants with available data were analyzed. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo 100 mg QD; EP547 100 mg QD | EP547 100 mg QD; EP547 100 mg QD
Number analyzed (Participants) | 27 | 25
scores on a scale | -3.7 (0.78) | -3.8 (0.82)

3. Secondary Outcome: Percentage of Participants With Improvement in Pruritus as Defined by Patient Global Impression of Change (PGI-C) at Week 6
Description: Participants were asked to rate their impression of overall change in pruritus in the past 7 days compared to before they started taking study drug using the PGI-C, a 7-point scale ranging from "much improved" to "much worse," with higher scores indicating less improvement in pruritus. Participants that reported a change in their itch of "minimally improved" or better were considered to be responders in terms of "improvement in pruritus."
Time Frame: Baseline; Week 6
Population: Full Analysis Set. Only participants with available data were analyzed. Exact binomial (Clopper-Pearson) confidence intervals have been reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo 100 mg QD; EP547 100 mg QD | EP547 100 mg QD; EP547 100 mg QD
Number analyzed (Participants) | 27 | 28
percentage of participants | 55.6 [35.3 to 74.5] | 60.7 [40.6 to 78.5]

4. Secondary Outcome: Percentage of Participants With Improvement in Pruritus Severity From Baseline as Defined by Change in Patient Global Impress of Severity (PGI-S) at Week 6
Description: Participants were asked to rate the severity of their pruritus in the past 7 days using the PGI-S, a 4-point scale ranging from "none" to "severe." Participants that reported a positive shift in their categorical assessment of itch compared to their Baseline level (e.g., "severe" at Visit 2 [Day 1] with a shift to "moderate" at Visit 6 [Week 6]) were considered to be responders in terms of "improvement in pruritus."
Time Frame: Baseline; Week 6
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo 100 mg QD; EP547 100 mg QD | EP547 100 mg QD; EP547 100 mg QD
Number analyzed (Participants) | 27 | 28
percentage of participants | 56.0 [34.9 to 75.6] | 52.0 [31.3 to 72.2]

5. Secondary Outcome: Percentage of Participants With a Reduction in WI-NRS Score ≥2 From Baseline at Week 6
Description: Participants were asked to rate the severity of their worst level of itching in the past 24 hours using the daily WI-NRS, an 11-point scale ranging from 0 (no itching) to 10 (worst itching imaginable). Itching severity scores collected via the WI-NRS have been categorized in the as mild (<4), moderate (≥4 to <7), or severe (≥7). The average WI-NRS score using the daily values from the week before the first dose of study drug (including the WI-NRS score captured on Study Day 1 of dosing) served as the Baseline score. A weekly score was determined based on the average of all available daily scores of the week.
Time Frame: Baseline; Week 6
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo 100 mg QD; EP547 100 mg QD | EP547 100 mg QD; EP547 100 mg QD
Number analyzed (Participants) | 28 | 28
percentage of participants | 44.4 [25.5 to 64.7] | 35.7 [18.6 to 55.9]

6. Secondary Outcome: Percentage of Participants With a Reduction in WI-NRS Score ≥3 From Baseline at Week 6
Description: as for outcome 5
Time Frame: Baseline; Week 6
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo 100 mg QD; EP547 100 mg QD | EP547 100 mg QD; EP547 100 mg QD
Number analyzed (Participants) | 28 | 28
percentage of participants | 37.0 [19.4 to 57.6] | 25.0 [10.7 to 44.9]

7. Secondary Outcome: Percentage of Participants With a Reduction in WI-NRS Score ≥4 From Baseline at Week 6
Description: as for outcome 5
Time Frame: Baseline; Week 6
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo 100 mg QD; EP547 100 mg QD | EP547 100 mg QD; EP547 100 mg QD
Number analyzed (Participants) | 28 | 28
percentage of participants | 37.0 [19.4 to 57.6] | 17.9 [6.1 to 36.9]

8. Secondary Outcome: Percentage of Participants With a WI-NRS Score <4 at Week 6
Description: as for outcome 5
Time Frame: Baseline; Week 6
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo 100 mg QD; EP547 100 mg QD | EP547 100 mg QD; EP547 100 mg QD
Number analyzed (Participants) | 28 | 28
percentage of participants | 42.9 [24.5 to 62.8] | 35.7 [18.6 to 55.9]

9. Secondary Outcome: Double-blind Treatment Period: Number of Participants With Any Treatment-emergent Adverse Event (TEAE), Any ≥Grade 3 TEAE, Any Related TEAE, and Any TEAE That Led to Discontinuation of Study Drug
Description: An adverse event (AE) is any untoward medical occurrence in a participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable or unintended sign (including a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product. TEAEs are AEs with an onset after the first dose of study drug or existing events that worsened after the first dose during the study. TEAEs were graded for severity (mild [Grade 1], moderate [Grade 2], severe [Grade 3], life threatening [Grade 4], death [Grade 5]) using Common Terminology Criteria for Adverse Events (CTCAE), version 5.0. The investigator assessed whether the TEAEs were related or unrelated to the study drug.
Time Frame: up to the end of Week 6
Population: Safety Analysis Set: All participants who were randomized and took at least 1 dose of randomized study drug. Analysis was based on the treatment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo 100 mg QD; EP547 100 mg QD | EP547 100 mg QD; EP547 100 mg QD
Number analyzed (Participants) | 30 | 31
Participants
  Any TEAE | 15 | 18
  Any ≥Grade 3 TEAE | 0 | 0
  Any related TEAE | 5 | 5
  Any TEAE that led to discontinuation of study drug | 0 | 0

10. Secondary Outcome: Open-label Extension Period: Number of Participants With Any TEAE, Any ≥Grade 3 TEAE, Any Related TEAE, and Any TEAE That Led to Discontinuation of Study Drug
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable or unintended sign (including a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product. TEAEs are AEs with an onset after the first dose of study drug or existing events that worsened after the first dose during the study. TEAEs were graded for severity (mild [Grade 1], moderate [Grade 2], severe [Grade 3], life threatening [Grade 4], death [Grade 5]) using CTCAE, version 5.0. The investigator assessed whether the TEAEs were related or unrelated to the study drug.
Time Frame: from the beginning of Week 7 up to Week 12
Population: Open-label Extension Analysis Set: all participants who completed the Double-Blind Treatment Period and received at least 1 dose of study drug in the Open-Label Extension Period
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo 100 mg QD; EP547 100 mg QD | EP547 100 mg QD; EP547 100 mg QD
Number analyzed (Participants) | 29 | 29
Participants
  Any TEAE | 16 | 15
  Any ≥Grade 3 TEAE | 2 | 0
  Any related TEAE | 5 | 2
  Any TEAE that led to discontinuation of study drug | 0 | 0

11. Secondary Outcome: Double-blind Treatment Period: Number of Participants With Any Serious TEAE, Any ≥Grade 3 Serious TEAE, Any Related Serious TEAE, and Any Serious TEAE That Led to Discontinuation of Study Drug
Description: TEAEs are AEs with an onset after the first dose of study drug or existing events that worsened after the first dose during the study. A serious TEAE is any untoward medical occurrence, that at any dose: results in death; is life threatening; requires hospital admission or prolongs hospitalization; results in persistent or significant disability or incapacity; is a congenital anomaly/birth defect; or is a medically significant event that, based on appropriate medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent one of the previously listed outcomes. Serious TEAEs were graded for severity (mild [Grade 1], moderate [Grade 2], severe [Grade 3], life threatening [Grade 4], death [Grade 5]) using CTCAE, version 5.0. The investigator assessed whether the serious TEAEs were related or unrelated to the study drug.
Time Frame: up to the end of Week 6
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo 100 mg QD; EP547 100 mg QD | EP547 100 mg QD; EP547 100 mg QD
Number analyzed (Participants) | 30 | 31
Participants
  Any serious TEAE | 0 | 0
  Any ≥Grade 3 serious TEAE | 0 | 0
  Any related serious TEAE | 0 | 0
  Any serious TEAE that led to discontinuation of study drug | 0 | 0

12. Secondary Outcome: Open-label Extension Period: Number of Participants With Any Serious TEAE, Any ≥Grade 3 Serious TEAE, Any Related Serious TEAE, and Any Serious TEAE That Led to Discontinuation of Study Drug
Description: as for outcome 11
Time Frame: from the beginning of Week 7 up to Week 12
Population: Open-label Extension Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo 100 mg QD; EP547 100 mg QD | EP547 100 mg QD; EP547 100 mg QD
Number analyzed (Participants) | 29 | 29
Participants
  Any serious TEAE | 1 | 0
  Any ≥Grade 3 serious TEAE | 1 | 0
  Any related serious TEAE | 0 | 0
  Any serious TEAE that led to discontinuation of study drug | 0 | 0

13. Secondary Outcome: Double-blind Treatment Period: Number of Participants With Any Treatment-emergent (TE) Adverse Event of Special Interest (AESI), Any ≥Grade 3 TE AESI, Any Related TE AESI, and Any TE AESI That Led to Discontinuation of Study Drug
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. TEAEs are AEs with an onset after the first dose of study drug or existing events that worsened after the first dose during the study. AESI were considered to be any clinically meaningful new, worsening from Baseline, or abnormal laboratory findings or symptoms suggestive of acute kidney injury (AKI) (e.g., "blood urea increased" or "protein urine present" AEs as identified by the Standardized Medical Dictionary for Regulatory Activities [MedDRA] Query [SMQ] "Acute renal failure"). TE AESIs were graded for severity (mild [Grade 1], moderate [Grade 2], severe [Grade 3], life threatening [Grade 4], death [Grade 5]) using CTCAE, version 5.0. The investigator assessed whether the AE AESIs were related or unrelated to the study drug.
Time Frame: up to the end of Week 6
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo 100 mg QD; EP547 100 mg QD | EP547 100 mg QD; EP547 100 mg QD
Number analyzed (Participants) | 30 | 31
Participants
  Any treatment-emergent (TE) AESI | 0 | 0
  Any ≥Grade 3 TE AESI | 0 | 0
  Any related TE AESI | 0 | 0
  Any TE AESI that led to discontinuation of study drug | 0 | 0

14. Secondary Outcome: Open-label Extension Period: Number of Participants With Any Treatment-emergent (TE) AESI, Any ≥Grade 3 TE AESI, Any Related TE AESI, and Any TE AESI That Led to Discontinuation of Study Drug
Description: as for outcome 13
Time Frame: from the beginning of Week 7 up to Week 12
Population: Open-label Extension Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo 100 mg QD; EP547 100 mg QD | EP547 100 mg QD; EP547 100 mg QD
Number analyzed (Participants) | 29 | 29
Participants
  Any TE AESI | 0 | 0
  Any ≥Grade 3 TE AESI | 0 | 0
  Any related TE AESI | 0 | 0
  Any TE AESI that led to discontinuation of study drug | 0 | 0

15. Secondary Outcome: Number of Participants With Any Clinically Meaningful Changes From Baseline in Clinically Meaningful in Clinical Laboratory Test Results
Description: Clinical laboratory test results included results for clinical hematology, chemistry, coagulation, and thyroid function parameters . The investigator determined if changes were clinically meaningful.
Time Frame: up to the end of Week 12
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo 100 mg QD; EP547 100 mg QD | EP547 100 mg QD; EP547 100 mg QD
Number analyzed (Participants) | 30 | 31
Participants | 3 | 0

16. Secondary Outcome: Number of Participants With Any Clinically Meaningful Changes From Baseline in Vital Sign Measurements
Description: Vital sign measurements included measurements for blood pressure, pulse rate, oxygen saturation, body temperature, and respiratory rate. The investigator determined if changes were clinically meaningful.
Time Frame: up to the end of Week 12
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo 100 mg QD; EP547 100 mg QD | EP547 100 mg QD; EP547 100 mg QD
Number analyzed (Participants) | 30 | 31
Participants | 0 | 1

17. Secondary Outcome: Number of Participants With Any Clinically Significant Changes From Baseline in Electrocardiogram (ECG) Parameters
Description: ECG parameters included heart rate, RR interval, PR interval, QRS duration, or QT interval. The investigator determined if changes were clinically significant.
Time Frame: up to the end of Week 12
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo 100 mg QD; EP547 100 mg QD | EP547 100 mg QD; EP547 100 mg QD
Number analyzed (Participants) | 30 | 31
Participants | 0 | 0

18. Secondary Outcome: Plasma Concentration of EP547 and Metabolites
Description: The lower level of quantitation = 0.01 micrograms per milliliter (µg/mL) for EP547 and 0.005 μg/mL for EP3583.
Time Frame: 1, 2, and 3 hours postdose on Day 1 and Week 3; predose on Weeks 1, 2, and 6
Population: Pharmokinetic Set: all participants who received at least 1 dose of EP547 and provided adequate blood samples for bioanalysis
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Placebo 100 mg QD; EP547 100 mg QD | EP547 100 mg QD; EP547 100 mg QD
Number analyzed (Participants) | 0 | 31
nanograms per milliliter (ng/mL)
  EP547: Day 1, 1 hour postdose: number analyzed (Participants) | 0 | 30
  EP547: Day 1, 1 hour postdose |  | 2661.0 (159.42)
  EP547: Day 1, 2 hours postdose: number analyzed (Participants) | 0 | 30
  EP547: Day 1, 2 hours postdose |  | 5197.7 (93.75)
  EP547: Day 1, 3 hours postdose: number analyzed (Participants) | 0 | 30
  EP547: Day 1, 3 hours postdose |  | 5698.4 (75.27)
  EP547: Week 1, predose: number analyzed (Participants) | 0 | 30
  EP547: Week 1, predose |  | 6267.9 (51.54)
  EP547: Week 2, predose: number analyzed (Participants) | 0 | 29
  EP547: Week 2, predose |  | 5786.5 (56.27)
  EP547: Week 3, predose: number analyzed (Participants) | 0 | 29
  EP547: Week 3, predose |  | 6617.4 (49.06)
  EP547: Week 3, 1 hour postdose: number analyzed (Participants) | 0 | 29
  EP547: Week 3, 1 hour postdose |  | 11709.4 (39.25)
  EP547: Week 3, 2 hours postdose: number analyzed (Participants) | 0 | 29
  EP547: Week 3, 2 hours postdose |  | 12012.7 (30.98)
  EP547: Week 3, 3 hours postdose: number analyzed (Participants) | 0 | 28
  EP547: Week 3, 3 hours postdose |  | 11909.4 (49.76)
  EP547: Week 6, predose: number analyzed (Participants) | 0 | 28
  EP547: Week 6, predose |  | 4947.6 (91.61)
  EP3583: Day 1, 1 hour postdose: number analyzed (Participants) | 0 | 30
  EP3583: Day 1, 1 hour postdose |  | 308.5 (160.23)
  EP3583: : Day 1, 2 hours postdose: number analyzed (Participants) | 0 | 30
  EP3583: : Day 1, 2 hours postdose |  | 796.1 (104.08)
  EP3583: : Day 1, 3 hours postdose: number analyzed (Participants) | 0 | 30
  EP3583: : Day 1, 3 hours postdose |  | 910.6 (90.22)
  EP3583: Week 1, predose: number analyzed (Participants) | 0 | 30
  EP3583: Week 1, predose |  | 952.1 (56.10)
  EP3583: Week 2, predose: number analyzed (Participants) | 0 | 29
  EP3583: Week 2, predose |  | 948.2 (61.73)
  EP3583: Week 3, predose: number analyzed (Participants) | 0 | 29
  EP3583: Week 3, predose |  | 1028.9 (64.53)
  EP3583: Week 3, 1 hour postdose: number analyzed (Participants) | 0 | 29
  EP3583: Week 3, 1 hour postdose |  | 1625.4 (54.57)
  EP3583: Week 3, 2 hours postdose: number analyzed (Participants) | 0 | 29
  EP3583: Week 3, 2 hours postdose |  | 1898.0 (47.98)
  EP3583: Week 3, 3 hours postdose: number analyzed (Participants) | 0 | 28
  EP3583: Week 3, 3 hours postdose |  | 1836.0 (62.20)
  EP3583: Week 6, predose: number analyzed (Participants) | 0 | 28
  EP3583: Week 6, predose |  | 801.8 (103.25)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: For participants who received placebo up to Week 6 and then switched to EP547, adverse events are presented by the treatment they were on at onset of the event.
Groups:
- Placebo: Participants were randomized to receive oral placebo 100 milligrams (mg) once daily (QD) for 6 weeks in the Double-Blind (DB) Treatment Period.
- EP547: Participants were randomized to receive oral EP547 100 mg QD for 6 weeks in the DB Treatment Period and for 6 weeks in the Open-Label Extension Period. Participants who were randomized to receive oral placebo 100 mg QD for 6 weeks during the DB Treatment Period received EP547 100 mg QD for 6 weeks in the Open-Label Extension Period.
Arm/Group | Placebo | EP547
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/30 | 1/60
Other Adverse Events (participants affected / at risk) | 7/30 | 24/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=30) | EP547 (N=60)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Gun shot wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=30) | EP547 (N=60)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 6 (6)
Headache (Nervous system disorders) | 3 (3) | 6 (15)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (5)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 4 (4)
Urinary tract infection (Infections and infestations) | 0 (0) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2023-10-02): https://cdn.clinicaltrials.gov/large-docs/20/NCT05525520/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-01): https://cdn.clinicaltrials.gov/large-docs/20/NCT05525520/SAP_001.pdf